CLINICAL TRIAL: NCT02164994
Title: Prospective Evaluation of the Long-term (18 Months) Effectiveness of the Femtosecond Laser-assisted Arcuate Incisions Following Cataract Surgery
Brief Title: Prospective Evaluation of the Long-term Effectiveness of the Femtosecond Laser-assisted Arcuate Incisions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 1402
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Astigmatism
Keywords: Astigmatism, arcuate incisions, astigmatic keratotomy
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical study is an open, controlled, prospective, single center, single-surgeon, post-market-clinical-follow-up study to evaluate the long-term (18 months) effectiveness of the femtolaser-assisted astigmatic keratotomy.

DETAILED DESCRIPTION:
The purpose of this prospective post-market-clinical-follow-up study is to address the long-term effectiveness of arcuate incisions, in eyes after VICTUS femtosecond laser-assisted astigmatic keratotomy.

This study will be conducted at Gemini eye clinic in Zlin, Czech Republic by Dr. Pavel Stodulka who will examine up to 100 eyes who previously received VICTUS femtolaser-assisted arcuate incisions treatment.

Patients will be recruited according to the study inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Clear corneal media
* Patients must be at least 40 years of age
* VICTUS™ femtosecond laser-assisted arcuate incisions surgery
* Preoperative Keratometric astigmatism: ≥ 1.0D and ≤ 3D
* Patients must have read, understood the Patient Information and signed the informed consent form
* Patients are willing and able to return for follow-up examinations

Exclusion Criteria:

* Corneal disease or pathology, such as corneal scaring
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Manifest Glaucoma
* Known sensitivity to planned concomitant medications
* Patients regularly taking medicines that could influence the result of the treatment respectively the vision
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Patients with keratoconus, keratectasia or other irregular cornea changes
* Patients with connective tissue weakness
* Subjects who are immune compromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, insulin dependent diabetes mellitus, autoimmune diseases, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis, collagenosis and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Abnormal examination results from slit lamp, fundus examination or IOLMaster; age related changes are acceptable
* Patients with eye diseases which decreases the visual acuity such as macular degeneration, macular edema, proliferative diabetic retinopathy
* Abnormal examination results from topography, age related changes are acceptable
* Patients who are pregnant or nursing
* Patients with concentration disorders, epilepsy and other complicating diseases
* Patients who are participating in another clinical study 30 days before

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only the patients who were previously treated with VICTUS™ femtosecond laser-assisted arcuate incisions and successfully pass the eligibility criteria are eligible for this follow-up extension study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative keratometric cylinder | 18 months after the VICTUS femtosecond laser-assisted arcuate incisions.
  Postoperative Astigmatism (keratometry) ≤ 1.0 D in 60% of eyes

SECONDARY OUTCOMES:
Postoperative Manifest Cylinder | 19 months after VICTUS femtosecond laser-assisted arcuate incisions treatment.
  Postoperative Manifest Astigmatism (manifest refraction) ≤ 1.0 D in 60% of eyes
Postoperative Objective Cylinder | 18 months after VICTUS femtosecond laser-assisted arcuate incisions treatment.
  Postoperative Objective Astigmatism (manifest refraction) ≤ 1.0 D in 60% of eyes

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, Dr. med, PhD, Principal Investigator — Gemini clinic, Zlin Pavel Stodulka, Dr. med Study Principal Investigator Gemini eye clinic
Locations (1):
- Gemini Eye Clinic, Zlín, Czechia